CLINICAL TRIAL: NCT00075816
Title: A Phase III Randomized, Multicenter Trial Comparing G-CSF Mobilized Peripheral Blood Stem Cell With Marrow Transplantation From Human Leukocyte Antigen (HLA) Compatible Unrelated Donors (BMT CTN #0201)
Brief Title: Peripheral Blood Stem Cell Transplant vs Bone Marrow Transplant in Individuals With Hematologic Cancers (BMT CTN 0201)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Blood and Marrow Transplant Clinical Trials Network (Network); National Cancer Institute (NCI) (NIH); National Marrow Donor Program (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BMTCTN0201; U01HL069294-05 (NIH); BMT CTN 0201 (Other: Blood and Marrow Transplant Clinical Trials Network); 5U24CA076518 (NIH); NCT00321776 (obsolete NCT alias); NCT00473395 (obsolete NCT alias)
Record Dates: First submitted 2004-01-09; First posted 2004-01-13 (Estimated); Results first posted 2016-02-01 (Estimated); Last update posted 2023-01-04 (Actual); Status verified 2022-12

CONDITIONS: Leukemia; Myeloproliferative Disorders; Myelodysplastic-Myeloproliferative Diseases
MeSH Terms: conditions — Leukemia; Myeloproliferative Disorders; Myelodysplastic-Myeloproliferative Diseases | interventions — Peripheral Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bone Marrow Transplant (Active Comparator): Allogeneic bone marrow transplantation
  Interventions: Biological: Allogeneic bone marrow transplantation
- Blood Stem Cell Transplant (Active Comparator): Peripheral blood stem cell transplantation
  Interventions: Biological: Peripheral blood stem cell transplantation

INTERVENTIONS:
Biological: Allogeneic bone marrow transplantation — Bone marrow transplant from HLA compatible unrelated donors.
  Arms: Bone Marrow Transplant
Biological: Peripheral blood stem cell transplantation — Peripheral blood transplant from HLA compatible unrelated donors.
  Arms: Blood Stem Cell Transplant

SUMMARY:
The study is designed as a Phase III, randomized, open label, multicenter, prospective, comparative trial of granulocyte colony stimulating factor (G-CSF)-mobilized peripheral blood stem cells (PBSC) versus marrow from unrelated donors for transplantation in patients with hematologic malignancies. Recipients will be stratified by transplant center and disease risk and will be randomized to either the PBSC or marrow arm in a 1:1 ratio.

DETAILED DESCRIPTION:
BACKGROUND:

Many studies of allogeneic marrow transplantation have shown that a higher dose of marrow cells correlates with more robust hematopoietic engraftment and lower mortality from infectious complications. Peripheral blood stem cells (PBSC) collected after mobilization with granulocyte colony stimulating factor (G-CSF) contain a larger number of CD34-positive (CD34) progenitors and total cells than bone marrow. These observations led to the hypothesis that transplantation of PBSC would lead to lower mortality compared to transplantation of marrow. In addition, PBSC grafts have a higher T cell content, predicting a possibly more powerful anti-leukemia effect. However, the higher T cell content of PBSC may also lead to increased incidence and severity of acute and chronic graft-versus-host disease (GVHD). This concern is especially serious when the donor is unrelated to the recipient. This prospective, randomized, multicenter clinical trial of unrelated donor transplantation will test the hypothesis that transplantation of PBSC leads to similar patient survival compared to transplantation of marrow.

DESIGN NARRATIVE:

This is a Phase III randomized, open label, multicenter clinical trial sponsored by the National Marrow Donor Program (NMDP) and the National Institutes of Health (NIH). The objective of the trial is to test the null hypothesis that there is no difference in overall survival after PBSC versus marrow transplants from HLA compatible unrelated donors. The study will compare G-CSF-mobilized PBSC transplantation with bone marrow transplantation from HLA-compatible unrelated donors for patients with leukemia, myelodysplastic or myeloproliferative syndromes. Conditioning and GVHD prophylaxis regimens will vary by center and within centers, however, the center must declare before randomization what regimens will be used for each patient. The primary endpoint of this trial is 2-year survival following randomization. Secondary analyses will consider neutrophil and platelet recovery, acute and chronic GVHD, time off all immunosuppressive therapy, relapse, infections, adverse events and immune reconstitution. The trial will include evaluation of patient and donor quality of life, composition of the graft, and immune reconstitution. Accrual is anticipated for 3 years with a follow-up period of 3 years.

ELIGIBILITY:
Patient Inclusion Criteria:

One of the following diagnoses:

* Acute myelogenous leukemia at the following stages: first remission, second remission, third or subsequent remission, or not in remission
* Acute lymphoblastic leukemia at the following stages: first remission, second remission, third or subsequent remission, or not in remission
* Chronic myelogenous leukemia at the following stages: chronic phase, accelerated phase, or blast phase
* Myelodysplastic syndromes (MDS) at the following stages: refractory anemia; refractory anemia with ringed sideroblasts; refractory cytopenia with multilineage dysplasia; refractory cytopenia with multilineage dysplasia and ringed sideroblasts; refractory anemia with excess blasts-1 (5-10% blasts); refractory anemia with excess blasts-2 (10-20% blasts); myelodysplastic syndrome, unclassified; or MDS associated with isolated del (5q)
* Myeloproliferative diseases: chronic myelomonocytic leukemia; agnogenic myeloid metaplasia with myelofibrosis (idiopathic myelofibrosis); juvenile myelomonocytic leukemia
* Therapy-related acute myelogenous leukemia (AML) or MDS with prior malignancy that has been in remission for at least 12 months. If the remission is less than 12 months, Medical Monitor or Protocol Chair approval is required for eligibility

Patient Exclusion Criteria:

* Prior allogeneic or autologous transplants using any hematopoietic stem cell source; patients with secondary malignancies who have had a prior autologous transplant will be eligible; the prior autologous transplant must have been performed for the primary malignancy (such as lymphoma) and must have occurred 12 or more months prior to enrollment
* Lymphoma (11% of 2001 NMDP transplants), other malignant disorders (6%), and non-malignant disorders (9%)

Donor Inclusion Criteria:

* Matched for HLA-A, B, and DRB1 antigens

  1. One antigen mismatch at HLA-A, B, or DRB1 is acceptable with or without mismatch at HLA-C
  2. Typing is by DNA techniques: intermediate resolution for A, B, and C, and high resolution for DRB1. HLA-C typing is mandatory but will not count in the match.
* Willing to undergo both bone marrow harvest and G-CSF administration with apheresis
* Willing to be randomly assigned to either marrow or PBSC collection
* Adequate peripheral venous access for leukapheresis or willing to undergo placement of a central catheter
* Donor center affiliation with NMDP
* Additional donor inclusion criteria can be found in the Donor Companion Manual

Donor Exclusion Criteria:

* Pregnant (positive serum β-HCG) or uninterruptible breastfeeding
* Known allergy to G-CSF or to E. Coli-derived recombinant protein products
* History of autoimmune disorders
* History of deep vein thrombosis or venous thromboembolism
* History of iritis or episcleritis
* History of serious adverse reaction to anesthesia
* Thrombocytopenia (platelets less than 150,000 per mcL) at baseline evaluation
* Current treatment with lithium
* Presence of sickle hemoglobin as demonstrated by appropriate testing such as hemoglobin electrophoresis
* Receiving experimental therapy or investigational agents

Max Age: 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 551 (Actual)
Dates: Start 2004-01; Primary Completion 2013-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Horowitz, MD, Study Director — Center for International Blood and Marrow Transplant Research
Locations (45):
- United States (39):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - City of Hope National Medical Center, Duarte, California
  - UCSD Cancer Center, La Jolla, California
  - University of California, San Francisco, San Francisco, California
  - Stanford Hospital and Clinics, Stanford, California
  - University of Florida College of Medicine (Shands), Gainesville, Florida
  - Emory University, Atlanta, Georgia
  - Loyola University, Maywood, Illinois
  - IBMT (Indiana Blood and Marrow Transplant) at St Francis Franciscan Health, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Kansas Hospital, Kansas City, Kansas
  - University of Maryland, Baltimore, Maryland
  - DFCI/Brigham & Women's, Boston, Massachusetts
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Washington University/Barnes Jewish Hospital, St Louis, Missouri
  - Washington University/St. Louis Children's Hospital, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Hackensack University Medical Center Cancer Center, Hackensack, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Cohen Children's Hospital, New Hyde Park, New York
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Ohio State/Arthur G. James Cancer Hospital, Columbus, Ohio
  - University of Oklahoma Medical Center, Oklahoma City, Oklahoma
  - Oregon Health & Science University (Peds), Portland, Oregon
  - Oregon Health Sciences University, Portland, Oregon
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - Vanderbilt University, Nashville, Tennessee
  - Baylor University Medical Center, Dallas, Texas
  - Baylor College of Medicine/The Methodist Hospital, Houston, Texas
  - University of Texas/MD Anderson CRC, Houston, Texas
  - Texas Transplant Institute, San Antonio, Texas
  - Utah BMT/Primary Children's Medical Center, Salt Lake City, Utah
  - Utah BMT/University of Utah Medical School, Salt Lake City, Utah
  - Virginia Commonwealth University MCV Hospitals, Richmond, Virginia
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
- Canada (6):
  - Tom Baker Cancer Centre, Calgary, Calgary, Alberta
  - Vancouver General Hospital, Vancouver, British Columbia
  - Hamilton Health Sciences - McMaster Site, Hamilton, Ontario
  - Ottawa Hospital, Ottawa, Ontario
  - University of Toronto, Princess Margaret Hospital, Toronto, Ontario
  - Queen Elizabeth II Health Sciences Centre - Halifax, Halifax

IPD SHARING:
Plan to Share IPD: Yes
Results will be published in a manuscript
Supporting Information: Study Protocol, ICF
Time Frame: Within 6 months of official study closure at participating sites.
Access Criteria: Available to the public
URL: https://biolincc.nhlbi.nih.gov/home/

REFERENCES:
- [Result] Anasetti C, Logan BR, Lee SJ, Waller EK, Weisdorf DJ, Wingard JR, Cutler CS, Westervelt P, Woolfrey A, Couban S, Ehninger G, Johnston L, Maziarz RT, Pulsipher MA, Porter DL, Mineishi S, McCarty JM, Khan SP, Anderlini P, Bensinger WI, Leitman SF, Rowley SD, Bredeson C, Carter SL, Horowitz MM, Confer DL; Blood and Marrow Transplant Clinical Trials Network. Peripheral-blood stem cells versus bone marrow from unrelated donors. N Engl J Med. 2012 Oct 18;367(16):1487-96. doi: 10.1056/NEJMoa1203517. PMID 23075175
- [Result] Foley B, Cooley S, Verneris MR, Curtsinger J, Luo X, Waller EK, Anasetti C, Weisdorf D, Miller JS. Human cytomegalovirus (CMV)-induced memory-like NKG2C(+) NK cells are transplantable and expand in vivo in response to recipient CMV antigen. J Immunol. 2012 Nov 15;189(10):5082-8. doi: 10.4049/jimmunol.1201964. Epub 2012 Oct 17. PMID 23077239
- [Result] Switzer GE, Bruce JG, Harrington D, Haagenson M, Drexler R, Foley A, Confer D, Bishop M, Anderlini P, Rowley S, Leitman SF, Anasetti C, Wingard JR. Health-related quality of life of bone marrow versus peripheral blood stem cell donors: a prespecified subgroup analysis from a phase III RCT-BMTCTN protocol 0201. Biol Blood Marrow Transplant. 2014 Jan;20(1):118-27. doi: 10.1016/j.bbmt.2013.10.024. Epub 2013 Nov 1. PMID 24184336
- [Result] Waller EK, Logan BR, Harris WA, Devine SM, Porter DL, Mineishi S, McCarty JM, Gonzalez CE, Spitzer TR, Krijanovski OI, Linenberger ML, Woolfrey A, Howard A, Wu J, Confer DL, Anasetti C. Improved survival after transplantation of more donor plasmacytoid dendritic or naive T cells from unrelated-donor marrow grafts: results from BMTCTN 0201. J Clin Oncol. 2014 Aug 1;32(22):2365-72. doi: 10.1200/JCO.2013.54.4577. Epub 2014 Jun 30. PMID 24982459
- [Result] Khera N, Majhail NS, Brazauskas R, Wang Z, He N, Aljurf MD, Akpek G, Atsuta Y, Beattie S, Bredeson CN, Burns LJ, Dalal JD, Freytes CO, Gupta V, Inamoto Y, Lazarus HM, LeMaistre CF, Steinberg A, Szwajcer D, Wingard JR, Wirk B, Wood WA, Joffe S, Hahn TE, Loberiza FR, Anasetti C, Horowitz MM, Lee SJ. Comparison of Characteristics and Outcomes of Trial Participants and Nonparticipants: Example of Blood and Marrow Transplant Clinical Trials Network 0201 Trial. Biol Blood Marrow Transplant. 2015 Oct;21(10):1815-22. doi: 10.1016/j.bbmt.2015.06.004. Epub 2015 Jun 11. PMID 26071866
- [Result] Young JH, Logan BR, Wu J, Wingard JR, Weisdorf DJ, Mudrick C, Knust K, Horowitz MM, Confer DL, Dubberke ER, Pergam SA, Marty FM, Strasfeld LM, Brown JWM, Langston AA, Schuster MG, Kaul DR, Martin SI, Anasetti C; Blood and Marrow Transplant Clinical Trials Network Trial 0201. Infections after Transplantation of Bone Marrow or Peripheral Blood Stem Cells from Unrelated Donors. Biol Blood Marrow Transplant. 2016 Feb;22(2):359-370. doi: 10.1016/j.bbmt.2015.09.013. Epub 2015 Sep 25. PMID 26409243
- [Result] Burns LJ, Logan BR, Chitphakdithai P, Miller JP, Drexler R, Spellman S, Switzer GE, Wingard JR, Anasetti C, Confer DL; Blood and Marrow Transplant Clinical Trials Network. Recovery of Unrelated Donors of Peripheral Blood Stem Cells versus Recovery of Unrelated Donors of Bone Marrow: A Prespecified Analysis from the Phase III Blood and Marrow Transplant Clinical Trials Network Protocol 0201. Biol Blood Marrow Transplant. 2016 Jun;22(6):1108-1116. doi: 10.1016/j.bbmt.2016.02.018. Epub 2016 Mar 21. PMID 27013014
- [Derived] Lee SJ, Logan B, Westervelt P, Cutler C, Woolfrey A, Khan SP, Waller EK, Maziarz RT, Wu J, Shaw BE, Confer D, Horowitz MM, Anasetti C. Comparison of Patient-Reported Outcomes in 5-Year Survivors Who Received Bone Marrow vs Peripheral Blood Unrelated Donor Transplantation: Long-term Follow-up of a Randomized Clinical Trial. JAMA Oncol. 2016 Dec 1;2(12):1583-1589. doi: 10.1001/jamaoncol.2016.2520. PMID 27532508

RESULTS

PARTICIPANT FLOW:
Groups:
- Bone Marrow: Patients who underwent transplantation of bone marrow from unrelated donors; all randomized patients were included in the primary, intention-to-treat analysis.
- Peripheral-Blood Stem Cells: Patients who underwent transplantation of peripheral-blood stem cells from unrelated donors; all randomized patients were included in the primary, intention-to-treat analysis.
Period: Overall Study
Arm/Group | Bone Marrow | Peripheral-Blood Stem Cells
Started | 278 | 273
Completed | 264 | 262
Not Completed | 14 | 11
Not completed — Did not undergo transplantation | 14 | 11

BASELINE CHARACTERISTICS:
Population: All randomized patients were included in primary, intention-to-treat analysis.
Groups:
- Bone Marrow: Bone marrow transplant from HLA compatible unrelated donors
- Peripheral-Blood Stem Cells: Peripheral blood stem cell transplant from HLA compatible unrelated donors
- Total: Total of all reporting groups
Arm/Group | Bone Marrow | Peripheral-Blood Stem Cells | Total
Number analyzed (Participants) | 278 | 273 | 551
Age, Customized [Number; unit: participants]
  0-10 years | 9 | 9 | 18
  11-20 years | 26 | 11 | 37
  21-30 years | 42 | 45 | 87
  31-40 years | 42 | 49 | 91
  41-50 years | 52 | 55 | 107
  51-60 years | 69 | 75 | 144
  >=61 years | 38 | 29 | 67
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 110 | 127 | 237
  Male | 168 | 146 | 314
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 13 | 23
  Not Hispanic or Latino | 258 | 244 | 502
  Unknown or Not Reported | 10 | 16 | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 4 | 4 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 12 | 10 | 22
  White | 250 | 248 | 498
  More than one race | 5 | 0 | 5
  Unknown or Not Reported | 6 | 11 | 17
Diagnosis [Number; unit: participants]
  Acute myeloid leukemia | 130 | 131 | 261
  Acute lymphoblastic leukemia | 61 | 56 | 117
  Chronic myeloid leukemia | 29 | 37 | 66
  Myelodysplastic syndrome | 52 | 41 | 93
  Chronic myelomonocytic leukemia | 4 | 4 | 8
  Myelofibrosis | 2 | 4 | 6
Karnofsky performance-status score [Number; unit: participants] — Assesses patient self-perceived global quality of life and functioning (excellent, very good, good, fair, poor), where 100 equals perfect quality of life.
  participants
    90-100% | 172 | 154 | 326
    <90% | 68 | 74 | 142
    Unknown | 38 | 45 | 83
Cytomegalovirus serologic testing [Number; unit: participants]
  Seropositivity for CMV | 142 | 123 | 265
  Seronegativity for CMV | 121 | 138 | 259
  Unknown | 15 | 12 | 27
Conditioning regimen [Number; unit: participants]
  Cyclophosphamide and total-body irradiation | 133 | 133 | 266
  Cyclophosphamide and busulfan | 90 | 75 | 165
  Fludarabine, busulfan, and antithymocyte globulin | 39 | 40 | 79
  Fludarabine and melphalan | 16 | 25 | 41
GVHD prophylaxis [Number; unit: participants]
  Cyclosporine and methotrexate | 67 | 59 | 126
  Tacrolimus and methotrexate | 183 | 196 | 379
  Other | 28 | 18 | 46
Transplantation patients [Number; unit: participants]
  Underwent transplantation | 264 | 262 | 526
  Did not undergo transplantation | 14 | 11 | 25
Antithymocyte globulin treatment [Number; unit: participants] — Data on antithymocyte globulin treatment was not collected for patients who did not undergo transplantation. Data were also missing for several patients who did undergo transplantation.
  participants
    Antithymocyte globulin treatment | 65 | 72 | 137
    No Antithymocyte globulin treatment | 193 | 183 | 376
    Unknown | 20 | 18 | 38
Number of donor mismatches at HLA-A, B, C, and DRB1 [Number; unit: participants] — Data on donor HLA mismatch were not collected for patients who did not undergo transplantation.
  participants
    0 | 200 | 209 | 409
    1 | 55 | 50 | 105
    2 | 7 | 3 | 10
    3 | 2 | 0 | 2
    Missing | 14 | 11 | 25
CD34+ cell dose per kilogram (x10^-6) [Median (Inter-Quartile Range); unit: cell dose per kilogram (x10^-6)] — Data on CD34+ cell dose were missing for 121 patients in the bone marrow group and 25 in the peripheral-blood group.
  cell dose per kilogram (x10^-6) | 2.75 [1.94 to 4.53] | 7.70 [5.43 to 11.28] | 5.23 [1.94 to 11.28]

OUTCOME MEASURES:

1. Primary Outcome: Two-year Overall Survival
Description: Overall survival rate at 2 years according to an intention-to-treat analysis.
Time Frame: Measured at 2 years
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Bone Marrow | Peripheral-Blood Stem Cells
Number analyzed (Participants) | 278 | 273
percentage of patients | 46 [40 to 52] | 51 [45 to 57]

2. Secondary Outcome: Neutrophil Engraftment
Time Frame: Measured at Day 28
Measure: Number; unit: percentage of patients
Arm/Group | Bone Marrow | Peripheral-Blood Stem Cells
Number analyzed (Participants) | 278 | 273
percentage of patients | 87 | 97

3. Secondary Outcome: Platelet Engraftment
Time Frame: Measured at Day 180
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Bone Marrow | Peripheral-Blood Stem Cells
Number analyzed (Participants) | 278 | 273
percentage of patients
  Platelet engraftment >20K from time of transplant | 85.8 [75.3 to 92.0] | 91.6 [78.9 to 96.8]
  Platelet engraftment >50K from time of transplant | 80.3 [70.3 to 87.2] | 86.7 [76.2 to 92.8]

4. Secondary Outcome: Graft Failure
Time Frame: Measured at 28 and 100 days
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Bone Marrow | Peripheral-Blood Stem Cells
Number analyzed (Participants) | 278 | 274
percentage of patients | 9 [6 to 13] | 3 [1 to 5]

5. Secondary Outcome: Extensive Chronic Graft-versus-host Disease (GVHD)
Time Frame: Measured at 730 days
Measure: Number (95% Confidence Interval); unit: percentage of patients
Groups:
- Bone Marrow: Patients who received transplantation of bone marrow from unrelated donors.
- Peripheral-Blood Stem Cells: Patients who received transplantation of peripheral-blood stem cells from unrelated donors.
Arm/Group | Bone Marrow | Peripheral-Blood Stem Cells
Number analyzed (Participants) | 278 | 273
percentage of patients | 32 [26 to 38] | 48 [42 to 54]

6. Secondary Outcome: Chronic GVHD
Time Frame: Measured at 2 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bone Marrow | Peripheral-Blood Stem Cells
Number analyzed (Participants) | 278 | 273
percentage of participants | 41 [34 to 48] | 53 [45 to 61]

7. Secondary Outcome: Relapse
Description: Analysis restricted to patients who received the transplant.
Time Frame: Measured at 2 years
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Bone Marrow | Peripheral-Blood Stem Cells
Number analyzed (Participants) | 264 | 262
percentage of patients | 28.9 [23.3 to 34.7] | 27.5 [22.1 to 33.2]

8. Secondary Outcome: Infections
Description: Number of infection reports per patient.
Time Frame: Measured at 1 and 2 years
Population: Analysis restricted to patients who received the transplant.
Measure: Number; unit: participants
Arm/Group | Bone Marrow | Peripheral-Blood Stem Cells
Number analyzed (Participants) | 264 | 262
participants
  0 infections | 49 | 68
  1 infection | 52 | 50
  2 infections | 46 | 48
  3 infections | 30 | 25
  4 infections | 26 | 17
  5 infections | 18 | 16
  6 infections | 11 | 8
  >6 infections | 32 | 30

9. Secondary Outcome: Grades III-V Unexpected Adverse Events
Time Frame: Measured by 2 years
Measure: Number; unit: participants
Arm/Group | Bone Marrow | Peripheral-Blood Stem Cells
Number analyzed (Participants) | 278 | 273
participants
  Pulmonary/dyspnea | 1 | 0
  Pericarditis with pericardial effusion | 1 | 0
  Myocardial infarction | 1 | 1
  Malignancy: skin squamous cell CA | 1 | 0
  Acute renal failure | 1 | 0
  R portal vein obstruction | 1 | 0
  Right side pulmonary embolus | 1 | 1
  Facial trauma - fractured L lamina | 1 | 0
  Pulmonary embolism | 1 | 1
  Blindness | 1 | 0
  Confusion | 1 | 0
  Intra-abdominal hemorrhage | 1 | 0
  Death | 1 | 0
  Altered mental status | 1 | 0
  Pneumonia | 1 | 0
  Vascular: pulmonary embolus | 0 | 1
  Sudden death | 0 | 1
  Hypertensive crisis | 0 | 1
  Elevated LFT S | 0 | 1
  Hemolytic transfusion reaction | 0 | 1
  Confusion, dehydration, hygroma | 0 | 1
  Respiratory decompensation | 0 | 1
  Retinal tear | 0 | 1
  Retinopathy both eyes | 0 | 1

10. Secondary Outcome: Acute GVHD Grade II-IV
Time Frame: 100 days, 180 days
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Bone Marrow | Peripheral-Blood Stem Cells
Number analyzed (Participants) | 278 | 273
percentage of patients
  100 days from transplantation | 45.6 [39.1 to 51.9] | 46.7 [40.2 to 53]
  180 days from transplantation | 50 [43.1 to 56.4] | 51 [44.2 to 57.4]

11. Secondary Outcome: Acute GVHD Grade III-IV
Time Frame: 100 days, 180 days
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Bone Marrow | Peripheral-Blood Stem Cells
Number analyzed (Participants) | 278 | 273
percentage of patients
  100 days from transplantation | 13.8 [9.9 to 18.2] | 16.4 [12.2 to 21.2]
  180 days from transplantation | 14.9 [10.9 to 19.6] | 18.8 [14.3 to 23.8]

12. Secondary Outcome: Current Immunosuppressive (IS) Free Survival
Description: This outcome measure takes into account subsequent immunosuppressive therapy that may occur following discontinuation of initial immunosuppressive therapy.
Time Frame: Measured at 2 years
Population: No data collected.
Arm/Group | Bone Marrow | Peripheral-Blood Stem Cells
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Immune Reconstitution
Time Frame: Measured at 100 days, 6 months, and 1 and 2 years
Population: No data collected
Arm/Group | Bone Marrow | Peripheral-Blood Stem Cells
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Donor Recovery of Baseline Complete Blood Count (CBC) and White Blood Cell Count (WBC) Differential
Time Frame: Measured at 1, 6, and 12 months
Population: No data collected
Arm/Group | Bone Marrow | Peripheral-Blood Stem Cells
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Donor Recovery to Baseline Toxicity Scores
Time Frame: Measured at 1, 6, and 12 months
Population: No data collected
Arm/Group | Bone Marrow | Peripheral-Blood Stem Cells
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: Donor Quality of Life
Time Frame: Measured at 1, 6, and 12 months
Population: No data collected
Arm/Group | Bone Marrow | Peripheral-Blood Stem Cells
Number analyzed (Participants) | 0 | 0

17. Secondary Outcome: Patient Quality of Life
Time Frame: Measured at baseline, 6 months, and 1, 2, and 5 years
Population: No data collected
Arm/Group | Bone Marrow | Peripheral-Blood Stem Cells
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 3-years post-transplant
Description: Serious adverse events are defined as events associated with death, life-threatening event, disability, congenital anomaly, required intervention to prevent permanent impairment or damage, hospitalization or other serious adverse event. Only unexpected adverse events are reported here.
Arm/Group | Bone Marrow | Peripheral-Blood Stem Cells
Serious Adverse Events (participants affected / at risk) | 13/260 | 10/261
Other Adverse Events (participants affected / at risk) | 0/260 | 0/261
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bone Marrow (N=260) | Peripheral-Blood Stem Cells (N=261)
Myocardial infarction (Cardiac disorders) | 0 | 1 (1)
Pericarditis (Cardiac disorders) | 1 (1) | 0
Blindness (Eye disorders) | 1 (1) | 0
Retinal tear (Eye disorders) | 0 | 1 (1)
Retinopathy (Eye disorders) | 0 | 1 (1)
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0
Death (General disorders) | 1 (1) | 0
Sudden death (General disorders) | 0 | 1 (1)
Portal vein occlusion (Hepatobiliary disorders) | 1 (1) | 0
Pneumonia (Infections and infestations) | 1 (1) | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 1 (1) | 0
Hepatic enzyme increased (Investigations) | 0 | 1 (1)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0
Confusional state (Psychiatric disorders) | 1 (1) | 0
Renal failure acute (Renal and urinary disorders) | 1 (1) | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Hypertensive crisis (Vascular disorders) | 0 | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2009-10-28): https://cdn.clinicaltrials.gov/large-docs/16/NCT00075816/Prot_SAP_ICF_000.pdf